CLINICAL TRIAL: NCT06950320
Title: Clinical Outcome of Electrical Auricular Vagal Stimulation in Patients With Stable Symptomatic Chronic Heart Failure
Brief Title: Clinical Outcome of Electrical Transcutaneous Auricular Vagal Stimulation in Patients With Stable Symptomatic Chronic Heart Failure
Acronym: COETAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Regina Patricia Schukro, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EK-No: 2033/2012; 2033/2012 (Registry Identifier: Ethics commitee Medical University of Vienna)
Record Dates: First submitted 2025-02-27; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Chronic Heart Failure
Keywords: auricular vagal stimulation; chronic heart failure; 6-minute walking test

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients received a placebo device which was a look-a-like, that stimulated only for 1h hour and then stopped. Patients in both groups were told that they will not feel the stimulation after a while, which might contribute to a better blinding between the groups.
  Interventions: Device: Placebo
- treatment group (Active Comparator): P-STIM (Biegler, Mauerbach, Austria) is a battery-operated micro-stimulation appliance weighing 5 grams, designed as a disposable product for a single use. P-STIM is placed behind the patient's ear and connected to stimulation needles (usually 3 needles) on the auricle. For the study, only one stimulation needle was needed. P-STIM offers regular therapy over several days. The appliance transmits low frequency electric pulses to exposed nerve endings. The built-in microchip creates periods of stimulation and rest, each lasting approximately 3 hours. Stimulation was performed with a frequency of 1Hz for 40min followed by a break of 20 min. After some time, the patient may feel as if the intensity of stimulation is decreasing. A decrease in the perceived intensity of stimulation may however be subjective and have no bearing on the effectiveness of the therapy.
  Interventions: Device: P-STIM (Biegler, Mauerbach, Austria) is a battery-operated micro-stimulation appliance

INTERVENTIONS:
Device: P-STIM (Biegler, Mauerbach, Austria) is a battery-operated micro-stimulation appliance — P-STIM (Biegler, Mauerbach, Austria) is a battery-operated micro-stimulation appliance weighing 5 grams, designed as a disposable product for a single use. P-STIM is placed behind the patient's ear and connected to stimulation needles (usually 3 needles) on the auricle. For the study, only one stimulation needle was needed. P-STIMTM offers regular therapy over several days. The appliance transmits low frequency electric pulses to exposed nerve endings. The built-in microchip creates periods of stimulation and rest, each lasting approximately 3 hours. Stimulation was performed with a frequency of 1Hz for 40min followed by a break of 20 min.
  Arms: treatment group
Device: Placebo — The placebo device is a look-a-like, that stimulates only for 1h hour and then stops.
  Arms: Placebo

SUMMARY:
This study aims to investigate whether electrical vagus nerve stimulation in the auricle has an impact on the clinical presentation of heart failure. The device used, P-STIM, is already successfully applied in pain therapy and angiology (peripheral arterial disease, PAD) and will also be tested against a placebo in this study.

In preliminary studies, acupuncture was shown to improve the 6-minute walking distance in heart failure patients (Kristen et al., 2010). The investigators assume that acupuncture and P-STIM have similar effects, and this study also aims to improve the 6-minute walking distance as its primary endpoint. Additional endpoints include LVEF (left ventricular ejection fraction), NYHA classification, inflammatory markers (e.g., CRP, pro-BNP), and patients' quality of life.

Study Design:

Patients will be randomly assigned to either the placebo or the verum group. They will receive treatment for five weeks (with the device being replaced weekly) and undergo a follow-up examination after four weeks.

At the beginning and during follow-up, Left ventricular ejection fraction (measured by cardiac ultrasound), inflammatory markers in the blood, NYHA classification, and quality of life (assessed by questionnaire) will be recorded. The primary endpoint, the 6-minute walking distance, will be measured at baseline, two weeks after the start of treatment, and at the follow-up examination.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure
* NYHA Classification II-III
* Stable medication since at least 1 months
* LVEF <40%
* Patients must be able to understand study conditions
* No exclusion criteria
* Signed informed consent 6.1.3 Exclusion criteria
* Any electrical auricular vagal stimulation treatment within 6 months prior to base line visit
* Participation in another clinical trial within 3 months prior to base line visit
* Ventricular tachyarrhythmia within 1 month prior to base line visit
* Psoriasis vulgaris
* Hemophilia
* Cardiac pace makers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
6-minutes walking distance test | before treatment randomization, study day 21, 35 days after randomization
  patients were asked to walk at comfortable speed for 6min in one of our hospital corridors (30m long), distance was assessed by a physician

SECONDARY OUTCOMES:
SF 36, quality of life | before treatment randomization, 35 days after treatment randomization
  The 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures.
  The possible score ranges from 0 to 100 points whereby 0 points represent the greatest possible limitation of health, while 100 points represent the absence of health restrictions.
adverse events | before treatment randomization, study day 21, 35 days after randomization
  An AE/ADE is any adverse change from the subject's baseline condition, i.e. any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease which is considered to be clinically relevant be the physician that occurs during the course of the, whether or not considered related to the medical device.
  Adverse event /ADE include:
  * Exacerbation of a pre-existing disease.
  * Increase in frequency or intensity of a pre-existing episodic disease or medical condition.
  * Disease or medical condition detected or diagnosed after treatment with the medical device even though it may have been present prior to the start of the clinical investigation.
  * Continuous persistent disease or symptoms present at baseline that worsen following the start of the clinical investigation.
  * Lack of efficacy in the acute treatment of a life-threatening disease.
  * Events considered by the investigator to be related to clinical investigation-mandated procedures.
blood concentration of TNF alpha | before treatment randomization, 35 days after treatment randomization
  blood samples will be collected before treatment randomization and at end of study, measurement will be in picogram/millilitre
blood concentration of Interleucin 6 (IL6) | before treatment randomization, 35 days after treatment randomization
  blood samples will be collected, measurement will be in nanogram/litre
blood concentration of C-reactive protein (CRP) | before treatment randomization, 35 days after treatment randomization
  blood samples will be collected, measurement will be in milligram/decilitre
blood concentration of NT-proBNP | before treatment randomization, 35 days after treatment randomization
  blood samples will be collected, measurement will be in picogram/mililitre
left ventricular ejection fraction | before treatment randomization, 35 days after treatment randomization
  left ventricular ejection fraction will be assessed by an experienced cardiologist via echocardiography and will be expressed as percentage of a normal value
NYHA | before treatment randomization, 35 days after treatment randomization
  New York Heart Association Classification, will be expressed in 4 stages Class I (Mild) No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea (shortness of breath). Class II (Mild) Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea. Class III (Moderate) Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV (Severe) Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased.
blood pressure | before treatment randomization, 35 days after treatment randomization
  blood pressure will be assessed non-invasively by a cardiologist and will be expressed as millimeter mercury
ST-elevation | before treatment randomization, 35 days after treatment randomization
  will be detected via electrocardiogram which was performed by a cardiologist

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Sator, MD, Professor, Study Director — Medical University of Vienna, Dept. of Pain Therapy; Regina Patricia Schukro, MD, Principal Investigator — Medical University of Vienna, Dept. of Anaesthesiology
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zijlstra FJ, van den Berg-de Lange I, Huygen FJ, Klein J. Anti-inflammatory actions of acupuncture. Mediators Inflamm. 2003 Apr;12(2):59-69. doi: 10.1080/0962935031000114943. PMID 12775355
- [Background] Schneider A, Streitberger K, Joos S. Acupuncture treatment in gastrointestinal diseases: a systematic review. World J Gastroenterol. 2007 Jul 7;13(25):3417-24. doi: 10.3748/wjg.v13.i25.3417. PMID 17659687
- [Background] Schwartz PJ, De Ferrari GM, Sanzo A, Landolina M, Rordorf R, Raineri C, Campana C, Revera M, Ajmone-Marsan N, Tavazzi L, Odero A. Long term vagal stimulation in patients with advanced heart failure: first experience in man. Eur J Heart Fail. 2008 Sep;10(9):884-91. doi: 10.1016/j.ejheart.2008.07.016. Epub 2008 Aug 28. PMID 18760668
- [Background] Kristen AV, Schuhmacher B, Strych K, Lossnitzer D, Friederich HC, Hilbel T, Haass M, Katus HA, Schneider A, Streitberger KM, Backs J. Acupuncture improves exercise tolerance of patients with heart failure: a placebo-controlled pilot study. Heart. 2010 Sep;96(17):1396-400. doi: 10.1136/hrt.2009.187930. Epub 2010 Jun 15. PMID 20554511
- [Background] Coats AJ. The "muscle hypothesis" of chronic heart failure. J Mol Cell Cardiol. 1996 Nov;28(11):2255-62. doi: 10.1006/jmcc.1996.0218. PMID 8938579
- [Background] Anand IS, Latini R, Florea VG, Kuskowski MA, Rector T, Masson S, Signorini S, Mocarelli P, Hester A, Glazer R, Cohn JN; Val-HeFT Investigators. C-reactive protein in heart failure: prognostic value and the effect of valsartan. Circulation. 2005 Sep 6;112(10):1428-34. doi: 10.1161/CIRCULATIONAHA.104.508465. Epub 2005 Aug 29. PMID 16129801
- [Background] Lainchbury JG, Troughton RW, Strangman KM, Frampton CM, Pilbrow A, Yandle TG, Hamid AK, Nicholls MG, Richards AM. N-terminal pro-B-type natriuretic peptide-guided treatment for chronic heart failure: results from the BATTLESCARRED (NT-proBNP-Assisted Treatment To Lessen Serial Cardiac Readmissions and Death) trial. J Am Coll Cardiol. 2009 Dec 29;55(1):53-60. doi: 10.1016/j.jacc.2009.02.095. PMID 20117364
- [Background] Mann DL. Inflammatory mediators and the failing heart: past, present, and the foreseeable future. Circ Res. 2002 Nov 29;91(11):988-98. doi: 10.1161/01.res.0000043825.01705.1b. PMID 12456484
- [Background] Lecour S, James RW. When are pro-inflammatory cytokines SAFE in heart failure? Eur Heart J. 2011 Mar;32(6):680-5. doi: 10.1093/eurheartj/ehq484. Epub 2011 Feb 7. PMID 21303780
- [Background] Gullestad L, Ueland T, Vinge LE, Finsen A, Yndestad A, Aukrust P. Inflammatory cytokines in heart failure: mediators and markers. Cardiology. 2012;122(1):23-35. doi: 10.1159/000338166. Epub 2012 Jun 12. PMID 22699305
- [Background] Pomerantz BJ, Reznikov LL, Harken AH, Dinarello CA. Inhibition of caspase 1 reduces human myocardial ischemic dysfunction via inhibition of IL-18 and IL-1beta. Proc Natl Acad Sci U S A. 2001 Feb 27;98(5):2871-6. doi: 10.1073/pnas.041611398. PMID 11226333
- [Background] Kapadia SR. Cytokines and heart failure. Cardiol Rev. 1999 Jul-Aug;7(4):196-206. doi: 10.1097/00045415-199907000-00011. PMID 10423671
- [Background] Damas JK, Gullestad L, Ueland T, Solum NO, Simonsen S, Froland SS, Aukrust P. CXC-chemokines, a new group of cytokines in congestive heart failure--possible role of platelets and monocytes. Cardiovasc Res. 2000 Jan 14;45(2):428-36. doi: 10.1016/s0008-6363(99)00262-x. PMID 10728363
- [Background] Aukrust P, Ueland T, Muller F, Andreassen AK, Nordoy I, Aas H, Kjekshus J, Simonsen S, Froland SS, Gullestad L. Elevated circulating levels of C-C chemokines in patients with congestive heart failure. Circulation. 1998 Mar 31;97(12):1136-43. doi: 10.1161/01.cir.97.12.1136. PMID 9537339
- [Background] Torre-Amione G, Kapadia S, Benedict C, Oral H, Young JB, Mann DL. Proinflammatory cytokine levels in patients with depressed left ventricular ejection fraction: a report from the Studies of Left Ventricular Dysfunction (SOLVD). J Am Coll Cardiol. 1996 Apr;27(5):1201-6. doi: 10.1016/0735-1097(95)00589-7. PMID 8609343
- [Background] Aukrust P, Ueland T, Lien E, Bendtzen K, Muller F, Andreassen AK, Nordoy I, Aass H, Espevik T, Simonsen S, Froland SS, Gullestad L. Cytokine network in congestive heart failure secondary to ischemic or idiopathic dilated cardiomyopathy. Am J Cardiol. 1999 Feb 1;83(3):376-82. doi: 10.1016/s0002-9149(98)00872-8. PMID 10072227
- [Background] Schwartz PJ, De Ferrari GM. Sympathetic-parasympathetic interaction in health and disease: abnormalities and relevance in heart failure. Heart Fail Rev. 2011 Mar;16(2):101-7. doi: 10.1007/s10741-010-9179-1. PMID 20577900
- [Background] Peuker ET, Filler TJ. The nerve supply of the human auricle. Clin Anat. 2002 Jan;15(1):35-7. doi: 10.1002/ca.1089. PMID 11835542
- Available data/document: Study Protocol — https://ethikkommission.meduniwien.ac.at — studyplan/studyprotocol/patient informed consent form/timeline are available on homepage of ethics committee of the medical university of Vienna

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT06950320/Prot_SAP_000.pdf